CLINICAL TRIAL: NCT04411212
Title: Granulocyte Colony-stimulating Factor and Platelet-rich Plasma Group in Patients With Recurrent Implantation Failure
Brief Title: G-CSF and PRP in Patients With Recurrent Implantation Failure
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riyadh Fertility and Reproductive Health center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: G-CSF and PRP in RIF
Record Dates: First submitted 2020-05-27; First posted 2020-06-02 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: Infertility,Female
Keywords: IVF; Platelet-rich plasma; Granulocyte colony-stimulating factor; Recurrent implantation failure
MeSH Terms: conditions — Infertility, Female | interventions — Granulocyte Colony-Stimulating Factor; Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Granulocyte colony-stimulating factor and platelet-rich plasma (Active Comparator)
  Interventions: Drug: Granulocyte colony-stimulating factor and platelet-rich plasma group
- Control group (Other)
  Interventions: Other: Control group

INTERVENTIONS:
Drug: Granulocyte colony-stimulating factor and platelet-rich plasma group — Antagonist protocol is used . Oocyte retrieval under transvaginal ultrasound guidance is performed 34 to 36 hours after HCG administration. Autologous platelet-rich plasma is prepared from the blood using the two step centrifuge process. Under ultrasound guidance and complete aseptic procedures, 1 ml of the PRP is infused inside the uterus while performing the mock embryo transfer. Moreover, G-CSF (Filgrastim®, 300μg/0.5ml) is injected subcutaneously. G-CSF is injected weekly until the 12th gestation week or negative pregnancy test.
  Arms: Granulocyte colony-stimulating factor and platelet-rich plasma
Other: Control group — Antagonist protocol is used . Oocyte retrieval under transvaginal ultrasound guidance is performed 34 to 36 hours after HCG administration. Mock embryo transfer is performed without injecting anything inside the uterus.
  Arms: Control group

SUMMARY:
The aim of this randomized controlled trial is to determine whether granulocyte colony-stimulating factor and platelet-rich plasma can be used to enhance the IVF-ET outcomes in patients with recurrent implantation failure

ELIGIBILITY:
Inclusion Criteria:

• Patients with history of three or more unsuccessful IVF-ET cycles with at least 2 good quality embryos transferred

Exclusion Criteria:

* Endometriosis
* Uterine anomalies
* Asherman syndrome

Ages: 1 Year to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 112 (Estimated)
Dates: Start 2020-05-28 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
Clinical pregnancy rate | Five weeks after embryo transfer
  Gestational sac detected by ultrasound examination

CONTACTS AND LOCATIONS:
Overall Officials: Usama M Fouda, Prof., Study Chair — Riyadh Fertility and Reproductive Health center
Locations (1):
- Riyadh Fertility and Reproductive Health center, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No